CLINICAL TRIAL: NCT03863236
Title: A Prospective Multicenter Randomized Study of Perioperative Oral Nutritional Support for Patients Having Surgery for Colon Cancer. Peri-Nutri
Brief Title: A Study of Perioperative Oral Nutritional Support for Patients Having Surgery for Colon Cancer, Peri-Nutri
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 235/2018
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Sarcopenia
Keywords: colon cancer, nutritional support, complications, mortality,
MeSH Terms: conditions — Colonic Neoplasms; Sarcopenia | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular diet (Active Comparator): The control group (group 1) will continue their regular diet.
  Interventions: Dietary Supplement: regular diet
- nutritional support Resource 2.5 (Active Comparator): The intervention group (group 2) will get preoperative nutritional support two weeks before the operation and the nutritional support will continue 10 days after the operation.
  Interventions: Dietary Supplement: nutritional support Resource 2.5

INTERVENTIONS:
Dietary Supplement: regular diet — The control group (group 1) will continue their regular diet.
  Arms: regular diet
Dietary Supplement: nutritional support Resource 2.5 — The intervention group (group 2) will get preoperative nutritional support (Resource 2.5 Compact/fibre combact) two weeks before the operation and the nutritional support will continue 10 days after the operation.
  Arms: nutritional support Resource 2.5

SUMMARY:
This is a multicenter, unblinded, randomized study. The aim of this study is to research whether preoperative and postoperative oral nutritional supplement (ONS) (Resource 2.5 Compact/fibre compact) used at least 2 weeks prior the surgery and 10 days after surgery can improve the nutritional status of a colon cancer patient and reduce number of complications. The aim is also to investigate whether the oral nutritional support can shorten the hospital stay and improve the patients´ quality of life. The aim is also to find out whether the oral nutritional support can reduce 90-day mortality and improve disease free and overall survival.

Consecutive patients diagnosed with primary adenocarcinoma of the colon who are considered for radical surgical procedure are enrolled in this study provided that the inclusion criteria are filled.

Patients in the intervention group start oral nutritional support (ONS)2 portions a day for about 2 weeks prior to the operation starting at the time of randomization and continue ONS 10 days after the operation. Control group will continue with their regular diet without ONS until the operation. Both groups keep a food diary for 4 days right after the randomization and both one month and three months after the operation to assess the energy and nutrient intakes.

Laboratory markers, NRS 2002, quality of life questionnaire, exercise questionnaire, bioelectrical impedance analysis (BIA) and handgrip strength as well as body composition on computer tomography scan are assessed prior to any treatment or supplement in order to estimate the patients' well-being and nutritional status prior to surgical operation. Laboratory parameters and QoL questionnaire are repeated right before the operation on admission to hospital as well as about 30 and 90 days after the operation in addition to BIA, handgrip strength to assess the effect of nutritional support. Data on complications, infections, length of stay in the hospital and mortality are collected.

Another arm in this research is to discover more information on biological markers in colon cancer and cancer related malnutrition thus providing targets for future treatment and prognostic predictors. Tissue samples are collected during this research at the surgery.

DETAILED DESCRIPTION:
The hypothesis in this study are:

1. Perioperative ONS decreases surgery related morbidity
2. Perioperative ONS increases the quality of life after surgery
3. Perioperative ONS decreases the length of stay in institutional care
4. Perioperative ONS decreases 90-day mortality and improve 5-year survival
5. Perioperative ONS benefits the patients to tolerate the adjuvant chemotherapy with less side effects
6. Perioperative ONS protects patients from postoperative nutritional depletion

Primary end point is to investigate whether the preoperative oral nutritional support decreases the number of complications during the 30-day follow up after the surgery. Secondary end points are to study the effect of oral nutritional support on quality of life after surgery, length of hospital stay, disease free and overall survival.

Randomization:

Patients having a surgery for adenocarcinoma of the colon are randomized on their preoperative visit in the outpatient clinic about 2-3 weeks prior to surgery.

The patients are randomized in two different groups according to NRS-2002 results. Both groups contain equal number of patients with normally nourished patients (NRS-2002 1-2) and malnourished patients by NRS 3 or more. NRS >5 patients are excluded (nutritional support is recommended before the surgery). The control group (group 1) will continue their regular diet. The study group (group 2) will get preoperative nutritional support two weeks before the operation and the nutritional support will continue 10 days after the operation. The control group will continue their regular diet after the operation.

Thus the randomization groups will be (total number of patients 318):

1. no oral nutritional support (control group) n=159
2. pre and postoperative oral nutritional support (intervention group) n=159

Preoperative assessment and data-collection:

All patients attending this study have a visit in the out-patient clinic 2-3 weeks prior the surgery. The height and weight are measured at the baseline. 3 and 6 months previous weights recalled by patient. ASA (The American Society of Anesthesiologists) classification is estimated by anesthesiologist. Whole body computer tomography is done to assess the possibility of metastases or locally spread cancer. Laboratory markers including total blood count, CRP (C-reactive protein) , creatinine, sodium, potassium, albumin, prealbumin, HbA1c, CEA (Carcinoembryonic antigen), transferrin and lipids (LDL, HDL, triglycerides) concentration are measured. History of smoking, alcohol consumption and other diseases and medications are recorded. NRS-2002 questionnaire is filled, as well as QoL- questionnaire and exercise questionnaire. Bioelectrical impedance analysis (InBody) and handgrip strength are measured.

Laboratory parameters, as described above, are measured at the time of randomization, at admission to hospital on the morning of surgery, leaving the hospital and about 1 and 3 months and 1,2 and 5 years after surgery. BMI, hand grip strength, bioelectrical impedance analysis are collected and the patients fill the QoL-questionnaire and exercise questionnaire at the same time points. The side effects of chemotherapy are monitored, as well as discontinuation of chemotherapy. Complication form will be filled when necessary.

Follow- up:

Follow-up will be same as other colon cancer patients. The follow.up will continue 5 years and the only difference is 3 month phone call. Patients will also fill exercise and quality of life forms and bioimpedance and handgrip strength will be measured.

First follow up visit after the surgery is at the outpatient clinic 1 month after the surgery. At that time patient is interviewed about recovery from surgery, patients who went to health care center to recover from surgery are asked about the length of stay and possible complications after leaving the hospital. The patients´ fill the 4-day food diary, exercise questionnaire and QoL questionnaire (RAND-36). The blood samples are taken. Bioelectrical impedance analysis and handgrip strength are measured as well.

Second follow up at 3 months after the surgery is by phone. Then the recovery from surgery is checked, as well as patients are asked to keep 4-day food diary. The blood samples are collected. Patients fill quality of life and exercise questionnaire.

Patients have CEA, hemoglobin, leucocyte count and thrombocyte count measured every 3 months until 2 years, and every 6 months until 5 months on a routine basis. Whole body CT scan is done in a year after the surgery. There are also follow up CT scans at the oncology clinic on patients who receive adjuvant therapy. They will be utilized for analysis on recovery from the sarcopenia and its effect on survival and toxicity of chemotherapy. There are routine hospital visits 1,2 and 5 years after the surgery. Laboratory parameters, BMI, bioelectrical impedance analysis and handgrip strength are measures at each visit. The patients fill the QoL questionnaire and exercise questionnaire also at each time points. charlson comorbidity index and who classification are also marked.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary colon adenocarcinoma
* Curative operation is possible
* Patient has a life expectancy of at least 12 months
* Patient signs the informed consent and agrees to attend all study visits

Exclusion Criteria:

* Recurrent colon adenocarcinoma
* Metastatic disease
* Cancer that will require multiorgan resection
* Pregnant or suspected pregnancy
* Patient with a comorbid illness or condition that would preclude the use of surgery (ASA 5).
* Patients with concurrent or previous malignant tumors within 5 years before the study enrollment
* Patient undergoing emergency procedures
* Dialysis
* Liver dysfunction, child pugh B or worse
* NRS score <2 or >5
* BMI under 18.5
* Weight loss 15% or more past 6 months
* Serum albumin less than 30 without liver or renal dysfunction
* Chronic malnutrition: short bowel syndrome, previous gastrectomy, pancreatic dysfunction
* Language barrier or other reasons why informed consent is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | complications are studied in every patients 30 days after operation
  Primary end point is to investigate whether the pre and postoperative oral nutritional support decreases the number of complications during the 30-day follow up after the surgery

SECONDARY OUTCOMES:
Nutrition and Quality of life | 5-year
  study the effect of oral nutritional support on quality of life after surgery (RAND-65 questionnaire)
Disease free and overall survival | 5-year
  study the effect of oral nutritional support on patients disease free and overall survival
90-day mortality | 90 days
  effect of nutritional support on 90-day mortality
Hospital stay | 90 days
  The aim is also to investigate whether the oral nutritional support can shorten the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Juha Saarnio, docent, Study Director — Oulun yliopisto
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aro R, Ohtonen P, Rautio T, Saarnio J, Makarainen E, Haivala R, Makinen MJ, Tuomisto A, Schwab U, Merilainen S. Perioperative oral nutritional support for patients diagnosed with primary colon adenocarcinoma undergoing radical surgical procedures -Peri-Nutri Trial: study protocol for a randomized controlled trial. BMC Nutr. 2022 Sep 2;8(1):89. doi: 10.1186/s40795-022-00591-y. PMID 36050804